CLINICAL TRIAL: NCT04090645
Title: A Humanitarian Device Exemption Treatment Protocol of TheraSphere for Treatment of Unresectable Primary or Unresectable Secondary Liver Cancer
Brief Title: TheraSphere & Treatment of Unresectable Primary or Unresectable Secondary Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TheraSphere
Record Dates: First submitted 2019-04-03; First posted 2019-09-16 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Liver, Cancer of, Non-Resectable

STUDY DESIGN:
Intervention Model Description: TheraSphere® consists of insoluble glass microspheres where Y-90 is an integral constituent of the glass. The mean sphere diameter ranges from 20 to 30 µm. Each milligram contains between 22,000 and 73,000 microspheres. TheraSphere® is supplied in 0.6 mL of sterile, pyrogen-free water contained in a 1.0 mL vee-bottom vial secured within a 12 mm clear acrylic vial shield. TheraSphere® is available in six activity sizes: 3 GBq (81 mCi), 5 GBq (135 mCi), 7 GBq (189 mCi), 10 GBq (270 mCi), 15 GBq (405 mCi) and 20 GBq (540 mCi).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TheraShere in treatment of primary & secondary liver carcinoma (Other): TheraSphere® is delivered into the liver tumor through a catheter placed into the hepatic artery. The hepatic artery provides the main blood supply to the tumor in the liver, whereas the portal vein supplies blood to normal liver parenchyma. TheraSphere® is embolized within the tumor and exerts a local beta radiation radiotherapeutic effect with a relatively limited concurrent injury to surrounding normal tissue.
  Interventions: Device: TheraSphere

INTERVENTIONS:
Device: TheraSphere — TheraSphere® is delivered into the liver tumor through a catheter placed into the hepatic artery. The hepatic artery provides the main blood supply to the tumor in the liver, whereas the portal vein supplies blood to normal liver parenchyma. TheraSphere® is embolized within the tumor and exerts a local beta radiation radiotherapeutic effect with a relatively limited concurrent injury to surrounding normal tissue.

SUMMARY:
Protocol Synopsis Title A Humanitarian Device Exemption Use Protocol of TheraSphere® For Treatment of Unresectable Primary or Secondary Liver Neoplasia

Supplier BTG International Canada Inc.

Type of Clinical Use Post-Marketing: TheraSphere® commercially distributed under HDE # 980006

Objectives • Provide supervised access to TheraSphere® therapy at this institution

* Evaluate response to treatment
* Evaluate toxicities and adverse experiences associated with TheraSphere® treatment
* Evaluate survival time

Number of Patients Up to 100 patients per year, expandable following completion of the first cohort.

Patients will be excluded: if they have pre-existing diarrhea/illness, or if they have a co-morbid disease or condition that would preclude safe delivery of TheraSphere® treatment and place the patient at undue risk.

Required Lab Parameters AST or ALT <5 times ULN For HCC: Bilirubin ≤ 2.0 mg/dl (unless segmental infusion is used) Negative pregnancy test in premenopausal women For other primary or secondary liver neoplasia, bilirubin levels specific to the primary or secondary liver neoplasia will be determined to confirm suitability for TheraSphere® treatment Negative pregnancy test in premenopausal women

Endpoints Provide TheraSphere® for patients who it is determined by their treating physicians and/or tumor board that the device is appropriate for the treatment of unresectable HCC in accordance with the FDA recommendation of use of a HUD within its approved indication or for the treatment of the patient's other primary or secondary liver neoplasia and is in accordance with the FDA recommendation of use of a HUD outside of its approved indication.

Evaluate SAE's associated with TheraSphere® treatment.

TheraSphere® Treatment: Suggested Table of Time and Events. TIME Pre-Treatment Evaluation First Treatment First Follow-up Visit Second Treatment3 Post-Treatment Follow-up3 EVENTS -30 to -5 Days Day 0 Day 21 - 42 Day 30 - 90 3 months

* 24 months

DETAILED DESCRIPTION:
Introduction

TheraSphere® TheraSphere® consists of insoluble glass microspheres where Y-90 is an integral constituent of the glass. The mean sphere diameter ranges from 20 to 30 µm. Each milligram contains between 22,000 and 73,000 microspheres. TheraSphere® is supplied in 0.6 mL of sterile, pyrogen-free water contained in a 1.0 mL vee-bottom vial secured within a 12 mm clear acrylic vial shield. TheraSphere® is available in six activity sizes: 3 GBq (81 mCi), 5 GBq (135 mCi), 7 GBq (189 mCi), 10 GBq (270 mCi), 15 GBq (405 mCi) and 20 GBq (540 mCi).

TheraSphere® is delivered into the liver tumor through a catheter placed into the hepatic artery. The hepatic artery provides the main blood supply to the tumor in the liver, whereas the portal vein supplies blood to normal liver parenchyma. TheraSphere® is embolized within the tumor and exerts a local beta radiation radiotherapeutic effect with relatively limited concurrent injury to surrounding normal tissue.

Contraindications

Please refer to the current Package Insert. In brief, the use of TheraSphere® is contraindicated in patients:

* For whom deposition to the gastrointestinal tract may not be corrected by angiographic techniques;
* Who show shunting of blood to the lungs that could result in delivery of greater than 16.5 mCi of Y-90 to the lungs in a single treatment;
* In whom hepatic artery catheterization is contraindicated;
* Who have severe liver dysfunction or pulmonary insufficiency; and
* Who present with complete occlusion of the main portal vein.

Warnings / Precautions Please refer to the current Package Insert for details.

Adverse Effects of the Device on Health Based on clinical and preclinical animal experience with TheraSphere® and other Y-90 microspheres, certain possible adverse reactions have been identified. A listing and discussion of these events can be found in the current Package Insert.

Rationale for Use Surgical resection of the affected portion of the liver offers the best chance for disease-free survival in patients with HCC. Unfortunately, most HCC patients present with disease that is not amenable to resection (multifocal disease) or have other medical contraindications to surgery (limited hepatic reserve related to advanced cirrhosis or chronic hepatitis). Fewer than 15%1 of hepatoma patients are suitable surgical candidates.

Toxicity in TheraSphere®-treated patients was acceptable. Radiation pneumonitis is a concern with hepatic-directed radiation treatment in hepatoma.

While CRC metastatic to the liver is considered Stage IV disease, advances in perioperative care, imaging and surgical techniques have supported development of liver-directed therapies which may be used alone, in combination with chemotherapy, or integrated with surgical approaches.

Tumor ablation techniques include thermal ablation (radiofrequency or laser induced), cryoablation and chemical ablation. Radiofrequency ablation appears promising but results have been inconsistent with recurrence rates of 10% to 50%.37 Further studies are required to better understand the optimal use of ablation in the treatment of CRC liver metastases.

Chemotherapy can be delivered directly to the liver via hepatic arterial infusion (HAI) or transarterial chemoembolization (TACE).

TACE delivers chemotherapy directly to hepatic tumors along with the administration of embolic material. T

Liver directed radiotherapy using external beam radiotherapy to the liver is limited by the higher sensitivity to radiation of normal liver parenchyma versus tumor and the subsequent risk of radiation induced liver disease.

Hepatic artery directed regional therapy is commonly performed in patients with unresectable, hepatic-predominant NETs.

Yttrium-90 microspheres (both resin [SIR-Spheres] and glass [TheraSphere®]) have been used in the treatment of patients with advanced hepatic metastatic NET since the US FDA availability of these devices in 2002 and 2000 respectively.

Comprehensive Clinical Evidence Summary Available upon request.

Purpose

Objective/Goal

There are no hypotheses to be tested in this treatment protocol which has the following objectives:

* Provide oversight to treatment with TheraSphere® to eligible patients with HCC of the liver who are not surgical resection candidates.
* Evaluate patient experience, toxicities and overall survival associated with TheraSphere® treatment.

This protocol allows multiple treatments with TheraSphere® that may be delivered on an outpatient basis. Patients may receive a single dose to the whole liver, lobar or segmental treatment delivered as a sequence of treatments approximately 30-90 days apart. The principal clinician, working with other medical team members in Radiation Oncology, Interventional Radiology, Medical Oncology, Hepatology, Transplant Surgery, Surgical Oncology and Nuclear Medicine, will develop a specific treatment plan for each patient, based upon the presenting condition of the patient, the vascular anatomy and the desired goal of treatment.

This HCC Treatment Protocol will contribute to increasing the knowledge base and clinical experience with TheraSphere® at this institution. The patient response to treatment and adverse experiences will be documented in accordance with standard institutional practice.

Treatment Protocol Design This is an observational treatment use protocol that will provide IRB oversight and documentation of the clinical experience of patients undergoing treatment for liver carcinoma using TheraSphere® under an HDE. Participation involves no investigational or research procedures. Patients will be followed for treatment-related adverse experiences for 30 days after each treatment. Survival experience will be monitored in accordance with institutional practices.

Data Analysis Data analysis will be limited to descriptive reports of the number and characteristics of the patients treated and their clinical and adverse event experiences.

Treatment An overview of the Primary or Secondary Liver Neoplasia Treatment Protocol, with recommended evaluations and follow-up schedule, is presented in Table 1, Page 6 of the Microsoft Word file on the CD (or see Section 3.2.4). The nature and timing of clinical follow-up is determined by the referring clinician, in accordance with the standards of care for oncology practice.

Synopsis of Protocol Patients will be screened and, if eligible, they will be asked to provide consent in accordance with IRB approval at this site. TheraSphere® treatment will be planned, the dose will be ordered and initial treatment scheduled. The physician and patient also will discuss and agree upon a plan for alternative treatment, should the patient be found ineligible for safe delivery of TheraSphere® treatment at the time of the final safety imaging studies. TheraSphere® treatment is performed in the outpatient setting.

Prior to initial treatment, a Tc-99m MAA scan will be performed using standard institutional practices. If there is an uncorrectable risk of flow to the gastrointestinal organs or risk of excessive shunting to the lungs, TheraSphere® treatment will not be administered and the patient will receive alternative or no treatment as previously defined in the treatment plan

Following treatment, patients will remain at the hospital under medical observation until the physician determines that they can safely be discharged to home (usually 2-6 hours). All patients will be evaluated 3-6 weeks post-treatment to assess clinical experience and adverse experiences. Subsequently, patient status will be followed via communication with the referring physician to determine disease status and survival.

Frequency of Visits Patients will have 1-2 outpatient visits for pre-treatment evaluation to determine initial eligibility to receive TheraSphere®, followed by a treatment visit for outpatient delivery of TheraSphere®, and at least 1 follow-up visit 3-6 weeks after initial treatment.

Catheters will be placed in the hepatic artery in the angiography suites. Depending on scheduling or equipment availability, the patient may be moved, with the catheter in place, from one location to the other for the diagnostic portion of the TheraSphere® planning, in accordance with institutional practice.

If more than one treatment is given, additional follow-up visits will occur after each treatment following institutional guidelines.

Subsequent follow-up contacts will be made with the referring physician. Patients will be asked to provide consent for medical record review after treatment.

No scheduled hospitalizations will be required, unless the physician determines that the patient should be admitted following treatment for management of a complication or adverse experience.

Pre-Treatment Evaluation The clinician will explain the procedure and treatment options to the patient and, if the patient wishes to proceed with treatment, the patient will indicate informed consent in accordance with hospital IRB requirements.

Pre-treatment evaluation will include the initial screening by history, physical examination, laboratory and diagnostic studies (hepatic angiography and Tc-99m MAA Scan). A treatment plan will be developed, dosage will be calculated and the TheraSphere® dose vial will be ordered from the manufacturer (Nordion).

Clinical and Laboratory Diagnostic Procedures

A history, physical examination and clinical interview will be completed. The diagnostic laboratory studies usually performed within 30 days of beginning TheraSphere® treatment are:

* Complete blood count with differential and platelet count
* Prothrombin Time/Partial Thromboplastin Time
* Serum Chemistry Panel, including: Electrolytes, BUN, AST, ALT, Creatinine, LDH, Glucose, Alkaline Phosphatase, Albumin and Total Bilirubin; Serum alphafetoprotein level (optional)

Diagnostic Imaging Studies

The following diagnostic radiographic studies may be performed:

* Chest X-Ray: Standard views of the chest may be taken (at discretion of physician)
* Computed Tomography Scanning of the Abdomen/Liver or Magnetic Resonance Imaging of the Abdomen/Liver
* Tc-99m MAA Scan

CT or MR scanning of the liver will be performed and the images used to calculate the appropriate liver volume for TheraSphere® dose determination. Reasonable attempts will be made to use the same imaging modality as that used for pre-treatment for all subsequent evaluations of the patient related to dose determination.

The dose is calculated as described below using the appropriate reference liver volume and mass. Dosimetric techniques for TheraSphere® are discussed in detail in the peer-reviewed literature.22-25

The imaging scan also is used to document the location and size of the hepatic lesion(s) and vascular anatomy (MRI only) where possible.

Prior to first TheraSphere® treatment, a Tc-99m MAA scan will be performed to obtain a preliminary assessment of hepatic infusion and any potential extrahepatic shunting or gastrointestinal flow. A discussion of the use of Tc-99m MAA scans can be found in the peer-reviewed literature.22,24 Lung Shunt Fraction will be determined as the ratio of total lung counts divided by total hepatic plus lung counts.

To be eligible to receive TheraSphere® treatment, the potential absorbed dose to the lungs must be <30 Gy (<16.5mCi of injected activity) per treatment. Any uncorrected detectable gastrointestinal flow is a contraindication to TheraSphere® treatment.

Treatment Planning The principal clinician or AU will formulate the initial treatment plan, indicating the number and sequence of planned TheraSphere® treatments. The clinician will assure that the patient understands the two-stage screening process that is necessary for this treatment procedure. The physician and patient will discuss and agree on a contingency treatment plan, including the option of no treatment, in the event that the patient is found ineligible to receive TheraSphere® after catheter placement. The Treatment Plan may be modified following initial treatment, based on clinical experience and patient response to treatment. Treatment of a second target tissue will be timed to occur within 30-90 days of initial TheraSphere® treatment.

Note: Patients whose treatment plan includes subsequent treatment with TheraSphere® must satisfy all applicable exclusion criteria again, prior to treatment.

TheraSphere® Dose Calculation (See Appendix 1 - Package Insert) The most commonly used target dose of TheraSphere®, within the approved dose range of 80-150 Gy, is 110-120 Gy. Depending on the timing of the product order relative to the TheraSphere® production schedule, and the treatment date proposed for the patient, it may be necessary to allow TheraSphere® to physically decay (see Table 3, TheraSphere® Package Insert, Appendix 1 of the Microsoft Word file on the CD) to the appropriate targeted activity before injection.

The amount of radioactivity required to deliver the dose to the selected liver target is calculated using the following formula:

Activity Required (GBq) = [Desired Dose (Gy)][ Mass of Selected Liver Target (kg)] 50

In nearly all cases, more than 95% of the glass microspheres are delivered. Calculation of the liver dose (Gy) delivered after injection uses the following formula:

Dose (Gy) = 50 [Injected Activity (GBq)][1-F][1-R] Mass of Selected Liver Target (kg)

where F is the fraction of injected activity deposited into the lungs as measured by Tc-99m MAA and R is the calculated residual.22

If there are questions, or if a follow-up contact is required, TheraSphere® Customer Support.

TheraSphere® is viable for therapeutic use for up to 12 days after the calibration date. TheraSphere® will be shipped by Nordion to ensure that TheraSphere® is on-site by the proposed treatment date. To meet the desired absorbed dose to the patient's liver, the clinician must schedule the patient's TheraSphere® treatment visit to occur within 12 days of the calibration date, and take into consideration the appropriate physical decay of the dose activity.

Procedures on Day of Treatment Treatment with TheraSphere® may be performed in the outpatient setting. The following sections describe the procedures performed on day of treatment.

Catheter Placement and TheraSphere® Infusion The goals of percutaneous catheter placement for TheraSphere® administration are: first, to limit the perfusion to the normal liver and, second, to deliver TheraSphere® as specified in the treatment plan.

On the day of treatment, TheraSphere® is administered via infusion under imaging guidance through an hepatic arterial catheter appropriately positioned in the arterial anatomy to permit selective infusion of TheraSphere® into the target tissue selected for treatment. The Interventional Radiologist will perform this procedure. The patency of the catheter will be maintained using standard techniques.

Administration of TheraSphere® The TheraSphere® administration procedure is described in the TheraSphere® Package Insert (Appendix 1) and in peer-reviewed literature.22-25

Patient Management Post-Treatment Care: Following treatment, the patient will remain under observation consistent with standard care guidelines for aftercare procedures involving arterial catheterization. T Supportive Care: Any concomitant medication or therapy deemed necessary to provide adequate supportive care to the patient in the post-treatment period will be administered according to institutional procedures.

Concurrent Treatments: In general, it is not recommended that patients receive other cancer therapy while receiving TheraSphere® treatment or within 4 weeks of completing the last TheraSphere® treatment plan. As the probability of adverse events is higher within first 30 days, this will facilitate assignment of cause.

Multiple Treatments with TheraSphere® If the patient's tumor distribution and hepatic arterial anatomy indicate that segmental or lobar treatment is appropriate, additional treatment procedures may be performed at approximately 4-12 week intervals until all tumors in the liver have been treated. At the time of pre-treatment evaluation, the principal clinician and collaborating physician(s) will formulate a treatment plan indicating whether a single or multiple treatment approach is to be implemented. This plan may be modified subsequently, based on the initial treatment experience.

The second treatment should occur not less than 30 days following the initial treatment. Prior to each treatment, the patient again must meet the inclusion/exclusion criteria as defined previously (Section 3.5.6).

Post-Treatment Follow-Up

Three- to Six-Week Follow-up Since the majority of microsphere radioactivity has decayed by 12 days, patients should be evaluated at 3-6 weeks post-treatment. The clinician can also evaluate the patient for a second treatment to the other lobe to be delivered at the appropriate time following the initial treatment.

Assess tumor response to the first infusion and overall clinical status of the patient. Tumor marker levels may increase, decrease or return to baseline at 30 days and due to this uncertainty, assessment of tumor markers should be reserved for long-term follow-up.

The following procedures may be performed at follow-up:

* Physical exam and clinical interview
* Solicitation and assessment of adverse events and adverse device effects
* Laboratory studies. The following laboratory studies may be repeated:
* Hematology: Complete blood count (CBC) with differential and platelet count
* Serum chemistry: Electrolytes, ALT, AST, alkaline phosphatase, BUN, LDH, creatinine, total bilirubin, albumin and glucose
* Tumor marker for HCC: Alpha-fetoprotein assay (AFP)
* Tumor marker(s) as appropriate for the other primary or secondary liver neoplasia being treated

Radiation Safety in the Post-Treatment Period If a patient receives a liver transplant or dies in the immediate period following treatment with TheraSphere®, radiation safety guidelines for handling of the body and/or body tissues should be followed, as dictated by institutional radiation safety policy.

Most patients have surface dose rates <20µSv/h at 30 days following treatment. Generally a patient skin surface dose rate of <20µSv/h does not require special handling (such as lead gloves, special instruments and extremity radiation monitors) by the surgeon during the operation. Notify radiation safety personnel for transportation and storage of the explanted tissue.

Device Dosages The target dose of TheraSphere® most commonly used is 120 Gy. Standard radiation safety techniques should be used.

Human Subjects Considerations

Potential Risks:

Exposure to Ionizing Radiation

Potential Risks of Radiation Exposure to the Patient

Potential Risks of Radiation Exposure to Attending Health Professionals

Risks of Hepatic Artery Catheterization

Blood Loss from Participation

Consent Procedures Informed consent is not a requirement for use of an HUD since use of an HUD does not constitute research or an investigation, which would normally require informed consent. Patient consent will be obtained in accordance to standard hospital practice.

Fully informed consent will be obtained by the principal clinician at the time of the initial referral consultation and documented in accordance with IRB requirements. The device and the protocol for treatment will be fully explained to the patient. The patient will have an opportunity to discuss the proposed treatment, including potential benefits and risks of the procedure, with his/her doctor before providing informed consent.

Protection of Subjects All patients will be under close supervision of the principal clinician for the duration of the treatment procedure and routinely following each treatment. Treatment planning and dose calculation will be performed in conjunction with the AU. Treatment will be delivered in an environment fully equipped to handle any medical emergencies occurring during treatment. No information will be published in a way that would identify any individual patient.

Confidentiality All screening studies and treatment procedures will be fully documented in the medical record according to institutional practice. The principal clinician will communicate with the referring physician regarding post-treatment outcomes. All results of treatment and communications with the referring physician will be kept strictly confidential. Clinical information will be released only with the expressed written consent of the patients except as may be required by law.

Potential Benefits to Subjects: Potentially Significant The clinical data suggest that this may be a suitable therapy for a disease with a particularly grim prognosis. With appropriate patient selection (see contraindications and warnings sections in Package Insert (Appendix 1) toxicities are low and survival data is promising (reports of >600 days in Okuda I patients15,16). ) Additional patient safety and outcome data are available for primary or secondary liver neoplasia in a number of cancer indications.

Risk-Benefit Ratio: Favorable The potential benefits to the patient participants may be significant. The ethics of providing this treatment have been assessed, at least in part, with the expectation that the treatment has the potential to provide direct benefits to patients and the treatment does not preclude them from subsequently receiving other standard alternative therapies for liver cancer.

Compensation No compensation or incentives will be provided to patients participating in this treatment.

Alternatives to Participation Alternatives to participation for patients with unresectable HCC or other liver cancer depend on the specifics of their neoplastic disease and general health status and may include systemic chemotherapy, liver transplantation, regional therapy using chemoembolization (CE) procedures and/or supportive care only. All of these other treatments may be provided to patients who have received TheraSphere® treatment. Due to the minimally embolic nature of TheraSphere®, the use of any other form of liver directed therapy is not precluded after TheraSphere® administration.

TheraSphere® is manfucatured by Nordion (Canada) Inc. for BTG International Canada Inc.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, of any race or sex, who have hepatocellular carcinoma of the liver, and who are able to give informed consent, will be eligible. Patients must have an ECOG Performance Status score of ≤ 2, with a life expectancy of ≥ 3 months, non-pregnant with an acceptable contraception in premenopausal women. Patients must be >4 weeks since prior radiation or prior surgery and at least 1 month post chemotherapy.

Exclusion Criteria:

* Contraindications to angiography and selective visceral catheterization

  * Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) per treatment of radiation to the lungs
  * Evidence of any detectable Tc-99m MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop or mitigate such flow (eg, placing catheter distal to gastric vessels)
  * Significant extrahepatic disease representing an imminent life-threatening outcome
  * Severe liver dysfunction or pulmonary insufficiency
  * Active uncontrolled infection
  * Significant underlying medical or psychiatric illness
  * Pregnancy

Patients will be excluded: if they have pre-existing diarrhea/illness, or if they have a co-morbid disease or condition that would preclude safe delivery of TheraSphere® treatment and place the patient at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Evaluate SAE's associated with TheraSphere® treatment | Day 21 after the first treatment till 24 months
  life saving measure_ days of survival after the treament

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Mantry, M.D., Principal Investigator — Methodist Health System
Locations (1):
- The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No